CLINICAL TRIAL: NCT05910580
Title: Improving Alcohol and Substance Use Care Access, Outcomes, and Equity During the Reproductive Years: A Type 1 Hybrid Trial in Family Planning Clinics
Brief Title: Improving Alcohol and Substance Use Care Access, Outcome, Equity During the Reproductive Years
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Stanford University (Other); Planned Parenthood League of Massachusetts (Other)
Responsible Party: Principal Investigator, Justine Welsh, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00005766; R01AA030529 (NIH)
Record Dates: First submitted 2023-05-19; First posted 2023-06-18 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Alcohol-Related Disorders; Substance-Related Disorders; Mental Health; Reproductive Health; Sexual Health; Sexually Transmitted Diseases; Contraception; Maternal Health; Pregnancy; Women's Health
Keywords: Implementation Science; Mass Screening; Motivational Interviewing; Referral and Consultation; Quality of Health Care; Early Medical Intervention; Family Planning Services; Primary Health Care; Reproductive Health Services; Telemedicine; Preconception Care; Young Adult
MeSH Terms: conditions — Alcohol-Related Disorders; Substance-Related Disorders; Psychological Well-Being; Sexually Transmitted Diseases | interventions — Mass Screening; Crisis Intervention

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Screening, Brief Intervention, and Referral to Treatment (SBIRT) (Experimental): Patients at study clinics who are randomized to receive the Screening, Brief Intervention, and Referral to Treatment (SBIRT) intervention, which is delivered in-person and through telemedicine.
  Interventions: Behavioral: Screening, Brief Intervention, and Referral to Treatment (SBIRT)
- Usual Care (No Intervention): Patients at study clinics who are randomized to receive usual care. None of the clinic sites have implemented standardized screening, brief intervention, or referral to treatment components. In this setting, usual care consists of basic quantity and frequency questions asked inconsistently as part of the admission process and varying by provider, with no standardized approach to screening, treatment, follow-up, or referral.

INTERVENTIONS:
Behavioral: Screening, Brief Intervention, and Referral to Treatment (SBIRT) — Screening, Brief Intervention, and Referral to Treatment (SBIRT) is an evidence-based approach supported by national healthcare organizations, including the Preventative Services Task Force and the American College of Obstetrics and Gynecologists. Validated tools will efficiently screen an individual's substance use risk. Patients who screen in the risky/harmful range then receive a brief motivational interviewing-based intervention adapted from the evidence-based Brief Negotiated Interview, lasting 5-10 minutes, which provides feedback, helps explore health risks, and motivates change. Individuals who screen in the severe category, indicating a likely AUD/SUD, also receive a brief intervention, aimed at increasing motivation to accept a referral to treatment, and requiring a more intensive approach will also receive a warm-hand off referral to specialty addiction treatment. Procedures for SBIRT delivery will be adapted to the flow of telemedicine visits.
  Arms: Screening, Brief Intervention, and Referral to Treatment (SBIRT)

SUMMARY:
The goal of this clinical trial is to test the effectiveness of evidence-based Screening, Brief Intervention, and Referral to Treatment (SBIRT) among adult patients who screen positive to one or more risky alcohol or substance use behaviors while seeking care at a sexual and reproductive health (SRH) clinic.

The main questions it aims to answer are:

* Does SBIRT impact patients' alcohol and substance use, SRH, mental health, physical health, quality of life, and wellbeing?
* Does SBIRT effectiveness differ by ethnicity, socioeconomic status, age, gender, and urbanicity?
* Does SBIRT effectiveness differ by delivery mode (in-person vs. telemedicine)?

Participants will receive in-person and telemedicine SBIRT, or usual care. Participants will complete surveys at interviews at baseline, 30 days, and 3 months.

Researchers will compare patients who received SBIRT to patients who receive usual care to see if patients who receive the SBIRT intervention have a greater reduction in negative outcomes as compared to those who receive usual care. In this setting, usual care consists of basic quantity and frequency questions asked inconsistently as part of the admission process and varying by provider, with no standardized approach to screening, treatment, follow-up, or referral.

DETAILED DESCRIPTION:
Risky alcohol and drug use are associated with severe, negative, and long-term health outcomes and disparities, including sexual and reproductive health (SRH), among reproductive aged people in the United States. High rates and sequelae of alcohol and drug use disproportionately experienced by structurally marginalized groups shape lifelong health inequities for people of racial/ethnic minority, living in poverty, and residing in under-resourced and under-served communities. Among populations at risk of pregnancy-related sequelae (predominantly those self-identifying as women and thus this study's primary focus), harmful alcohol and substance use and alcohol use disorders (AUDs)/substance use disorders (SUDs) contribute to condom and contraceptive nonuse among those not intending pregnancy, sex while intoxicated, non-consensual sex, violence/rape, sexually transmitted infections, unintended pregnancy, and maternal and infant morbidity and mortality.

Family planning (FP) clinics are uniquely well-suited but entirely untapped sites for implementing and scaling integrated alcohol/substance use services. Largely community-based health centers that are publicly funded and/or serve Medicaid enrollees, FP clinics are a trusted care source and primary access point for reproductive aged women, and a safety net for the most socially disadvantaged groups. Yet few, if any, studies have rigorously evaluated interventions or implementation strategies to accelerate the uptake of alcohol/substance services in FP contexts. In obstetrics and HIV, widespread adoption of evidence-based SBIRT (screening, brief intervention, and referral to treatment) is precluded by multi-level barriers; data on specific challenges faced by FP providers are lacking. Virtually nothing is known about telemedicine, which has been rolled out for contraception and other routine visits during the pandemic, as a technological infrastructure for SBIRT. Whether and how the promising strategy of Implementation and Sustainment Facilitation (ISF) can bridge systems barriers and support scale up in FP settings is unknown.

The researchers of this study propose an explanatory, sequential, mixed methods study of alcohol and drug SBIRT in an expansive FP clinic network - a novel and highly impactful setting with a national reach of a diverse and largely structurally disadvantaged population of reproductive-aged women at greatest risk for AUDs/SUDs. The researchers will conduct a randomized Type 1 Hybrid Effectiveness-Implementation Trial within a large Northeastern regional affiliate and its four clinics of a national SRH care organization.

Results will inform an evidence-based, innovative, stakeholder-driven FP SBIRT model in response to the high-level calls for integrated women's health care. With concrete guidance for scaling alcohol/ drug services in SRH settings nationally, findings will promote women's health equity across the U.S.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 years
* U.S. residing
* Have internet access (own a computer or smart phone)
* Screen positive to one or more risky alcohol and substance use behaviors as determined by our standardized abbreviated instruments

Exclusion Criteria:

* Not capable of communicating (reading, speaking, writing) in English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Average Number of Drinks Per Drinking Day | Baseline, Day 30, Month 3
  Participants are asked to self-report the number of drinks consumed on days when alcohol was consumed, during the past 30 days.
Number of Days of Drug Use | Baseline, Day 30, Month 3
  Participants are asked to self-report the number of days of drug use in the past 30 days.
Incidence of sex under influence of alcohol/drugs | Baseline, Day 30, Month 3
  Any incidence of sex under influence of alcohol/drugs in past 30 days.
Number of events of sex under influence of alcohol/drugs | Baseline, Day 30, Month 3
  The number of events of sex while under influence of alcohol/drugs in past 30 days.
Patient Health Questionnaire (PHQ-9) | Baseline, Day 30, Month 3
  The Patient Health Questionnaire (PHQ-9) is a 9-item instrument assessing symptoms of depression during the prior two weeks. Responses are given on a 4-point scale where 0 = not at all and 3 = nearly everyday. Total scores range from 0 to 27 where higher scores indicate greater feelings of depression. Scores of 0 to 4 indicate minimal depression, scores of 5 to 9 indicate mild depression, scores of 10 to 14 indicate moderate depression, scores of 15 to 19 indicate moderately severe depression, and scores of 20 or more indicate severe depression.
Number of Clinic Patients Receiving a Brief Intervention During Implementation Phase | During the 12-month implementation phase
  The number of patients in each clinic who screen positive receiving a brief intervention during the implementation phase of the study.
Number of Clinic Patients Receiving a Brief Intervention During Sustainment Phase | During the 12-month sustainment phase
  The number of patients in each clinic who screen positive who receive a brief intervention during the sustainment phase of the study.
Number of Providers Using SBIRT During Implementation Phase | During the 12-month implementation phase
  The number of providers in each clinic using SBIRT during the implementation phase.
Number of Clinics Using SBIRT During Sustainment Phase | During the 12-month sustainment phase
  The number of clinics using SBIRT during the sustainment phase.
Number of Providers Using SBIRT During Sustainment Phase | During the 12-month sustainment phase
  The number of providers in each clinic using SBIRT during the sustainment phase.
Number of Completed BIOS Tracking Sheets to Achieve Competency | During the preparation phase
  The number of completed Brief Intervention Observation Sheets (BIOS) needed to achieve competency will be examined.
Brief Intervention Observation Sheet (BIOS) Score | During the 12-month implementation phase
  Fidelity to the intervention is assessed as the mean score on the first 10 items of the Brief Intervention Observation Sheet (BIOS). The score per provider is determined from a sample of audio recorded brief interventions. Responses to items are recorded as a "yes" or "no" assessment of whether the steps of the brief intervention were completed. The total score is the number of "yes" items and can range from 0 to 10, with higher scores indicating more steps completed.
Brief Intervention Observation Sheet (BIOS) Score - Motivational Style | During the 12-month implementation phase
  Fidelity to the intervention is assessed as the mean score on the 11th item of the Brief Intervention Observation Sheet (BIOS). The score per provider is determined from a sample of audio recorded brief interventions. Item 11 assesses the overall motivational interviewing style used by the provider. Scores are rated on a 7-point scale where 1 = not at all and 7 = very effectively. Higher scores indicate greater motivational interviewing style.

SECONDARY OUTCOMES:
Number of Days of Alcohol Use | Baseline, Day 30, Month 3
  Participants are asked to self-report the number of days they consumed alcohol during the past 30 days.
Number of Days of Binge Drinking | Baseline, Day 30, Month 3
  Participants are asked to self-report the number of days they consumed 4 or more alcoholic drinks per day during the past 30 days.
Alcohol Use Disorders Identification Test-Concise (AUDIT-C) Score | Baseline, Day 30, Month 3
  The Alcohol Use Disorders Identification Test-Concise (AUDIT-C) is a 3-item alcohol screening instrument that reliably identifies persons who are hazardous drinkers or have active alcohol use disorders (including alcohol abuse or dependence). The questionnaire asks about drinking behavior in the past 30 days. Responses to items are given on a 5-point scale where 0 = never and 4 = the highest frequency of alcohol use or consumption per drinking day. Total scores range from 0 (non-drinkers) to 12. Higher scores indicate that a person's alcohol consumption is likely to affect his or her health and safety.
Drug Abuse Screening Test (DAST-10) Score | Baseline, Day 30, Month 3
  The Drug Abuse Screening Test (DAST-10) is a 10-item instrument assessing drug use (not including alcohol and tobacco use). Each item is responded to as "yes" or "no" and the total score is the sum of all "yes" responses. Total scores range from 0 to 10 with a score of 0 indicating that no problems are reported and the degree of problems related to drug abuse increase as the total score increases. Scores of 1 or 2 indicate a low level of problems, scores of 3 to 5 indicate a moderate level of problems, scores of 6 to8 indicate substantial levels of problems, and scores of 9 and 10 indicate severe levels of problems related to drug abuse.
Incidence of condom nonuse | Baseline, Day 30, Month 3
  Participants are asked to report any incidence of condom nonuse monogamous encounters in the past 30 days, among women not intending pregnancy.
Number of events of condom nonuse | Baseline, Day 30, Month 3
  Participants reporting condom nonuse are asked to report the number of events of condom nonuse monogamous encounters in the past 30 days, among women not intending pregnancy.
Incidence of contraceptive nonuse | Baseline, Day 30, Month 3
  Participants are asked to report any incidence of contraceptive nonuse monogamous encounters in the past 30 days, among women not intending pregnancy.
Number of events of contraceptive nonuse | Baseline, Day 30, Month 3
  Participants reporting contraception nonuse are asked to report the number of events of contraceptive nonuse monogamous encounters in the past 30 days, among women not intending pregnancy.
Incidence of regretted/nonconsensual sex and sexual violence | Baseline, Day 30, Month 3
  Participants are asked to report any incidence of non-consensual sex, regretted sex, or sexual violence in past 30 days.
Number of events of regretted/nonconsensual sex and sexual violence | Baseline, Day 30, Month 3
  Participants reporting non-consensual sex, regretted sex, or sexual violence in past 30 days are asked to report the number of events.
Unintended pregnancy | Baseline, Day 30, Month 3
  Participants are asked to report any incidence of unintended pregnancy occurring in the past 30 days.
Generalized Anxiety Disorder 7-item (GAD-7) Scale Score | Baseline, Day 30, Month 3
  The Generalized Anxiety Disorder 7-item (GAD-7) instrument is a well-validated patient self-report scale measuring anxiety severity. Participants respond to statements to indicate how often they have been bothered by specified symptoms of anxiety (such as "feeling nervous, anxious, or on edge). Response choices include 0 = not at all sure, 1 = several days, 2 = over half the days, and 3 = nearly every day. Total scores range from 0 to 21 with higher scores indicating increased anxiety. A score of 0 to 4 indicates minimal anxiety, scores of 5 to 9 indicate mild anxiety, scores of 10 to 14 indicate moderate anxiety, and scores of 15 to 21 indicate severe anxiety.
World Health Organization-Five Well-Being Index (WHO-5) Score | Baseline, Day 30, Month 3
  The World Health Organization-Five Well-Being Index (WHO-5) a 5-item scale that measures subjective psychological well-being in past 14 days. Responses to items are given on a 6-point scale where 0 = at no time and 5 = all of the time. Total raw scores range from 0 to 25, with 0 representing the worst possible and 25 representing the best possible quality of life. Scores can also be multiplied by 4 to obtain a percentage score ranging from 0 to 100, where 0 represents the worst possible quality of life and 100 represents the best possible quality of life.
General Self-reported Health Score | Baseline, Day 30, Month 3
  Likert rating of general self-reported health in past 30 days
12-Item Short Form (SF-12) Health Survey Score | Baseline, Day 30, Month 3
  Quality of life is assessed with the SF-12 Health Survey. The SF-12 is a multipurpose, standardized self-report short form survey with 12 questions assessing mental and physical functioning. The SF-12 consists of 12 items with a Likert-type response format that measures quality of life with a Physical Component Summary (PCS) and Mental Component Summary (MCS). Subscales associated with the PCS include physical functioning, role limitations due to physical problems, bodily pain, and general health perceptions. Subscales associated with the MCS include vitality (energy and fatigue), social functioning, role limitations due to emotional problems, and mental health. A scoring algorithm is used to generate a total score for each component ranging from 0 to 100. Low values represent a poor health state while high values represent a good health state.
Number of Patients Screened During Implementation Phase | During the 12-month implementation phase
  The number of patients, out of all patients seen at the study sites, who are screened during the implementation phase.
Number of Patients Screened During Sustainment Phase | During the 12-month sustainment phase
  The number of patients, out of all patients seen at the study sites, who are screened during the sustainment phase.
Number of Patients Receiving Referral During Implementation Phase | During the 12-month implementation phase
  The number of patients who screen at a severe level of alcohol use, who receive a referral during the implementation phase.
Number of Patients Receiving Referral During Sustainment Phase | During the 12-month sustainment phase
  The number of patients who screen at a severe level of alcohol use, who receive a referral during the sustainment phase.
University of Missouri-Kansas City Screening & Brief Intervention Knowledge Assessment Score | During the implementation phase
  SBIRT knowledge is assessed with the University of Missouri-Kansas City Screening & Brief Intervention Knowledge Assessment. This instrument will be completed by providers undergoing training in SBIRT. Scores range from 0-20, with higher scores indicating more knowledge of SBIRT.
Brief Intervention Observation Sheet (BIOS) Score During Preparation Phase | During the preparation and implementation phases
  Fidelity to the intervention is assessed as the mean score on the first 10 items of the Brief Intervention Observation Sheet (BIOS), from the last observation conducted during provider training. The score per provider is determined from a sample of audio recorded brief interventions. Responses to items are recorded as a "yes" or "no" assessment of whether the steps of the brief intervention were completed. The total score is the number of "yes" items and can range from 0 to 10, with higher scores indicating more steps completed.
Brief Intervention Observation Sheet (BIOS) Score - Motivational Style | During the preparation and implementation phases
  Fidelity to the intervention is assessed as the mean score on the 11th item of the Brief Intervention Observation Sheet (BIOS), from the last observation conducted during provider training. The score per provider is determined from a sample of audio recorded brief interventions. Item 11 assesses the overall motivational interviewing style used by the provider. Scores are rated on a 7-point scale where 1 = not at all and 7 = very effectively. Higher scores indicate greater motivational interviewing style.

OTHER OUTCOMES:
Number of Participants with STI Diagnosis | Baseline, Day 30, Month 3
  The number of participants receiving a diagnosis of one more sexually transmitted infections (STIs) in past 30 days.
Past or current receipt of substance use treatment or services | Baseline, Day 30, Month 3
  Number of days/times the participant received treatment or counseling for alcohol or drugs or attended a self-help/mutual support meeting in past 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Kelli S Hall, MD, Principal Investigator — Columbia University; Justine Welsh, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Greater Boston Health Center, Boston, Massachusetts
  - Metro West Health Center, Marlborough, Massachusetts
  - Western Massachusetts Health Center, Springfield, Massachusetts
  - Central Massachusetts Health Center, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Per the NIAAA Exemption Request Committee's determination electronic health records/administrative records data components will not be shared. Quantitative survey data will be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available for sharing following publication of finding from this study and will be available indefinitely.
Access Criteria: Anyone who wishes to access the data will be able to do so.

REFERENCES:
- [Background] Tan CH, Denny CH, Cheal NE, Sniezek JE, Kanny D. Alcohol use and binge drinking among women of childbearing age - United States, 2011-2013. MMWR Morb Mortal Wkly Rep. 2015 Sep 25;64(37):1042-6. doi: 10.15585/mmwr.mm6437a3. PMID 26401713
- [Background] Naimi TS, Lipscomb LE, Brewer RD, Gilbert BC. Binge drinking in the preconception period and the risk of unintended pregnancy: implications for women and their children. Pediatrics. 2003 May;111(5 Pt 2):1136-41. PMID 12728126
- [Background] Thomas AG, Brodine SK, Shaffer R, Shafer MA, Boyer CB, Putnam S, Schachter J. Chlamydial infection and unplanned pregnancy in women with ready access to health care. Obstet Gynecol. 2001 Dec;98(6):1117-23. PMID 11755563
- [Background] Kesmodel U, Wisborg K, Olsen SF, Henriksen TB, Secher NJ. Moderate alcohol intake in pregnancy and the risk of spontaneous abortion. Alcohol Alcohol. 2002 Jan-Feb;37(1):87-92. doi: 10.1093/alcalc/37.1.87. PMID 11825863
- [Background] Iyasu S, Randall LL, Welty TK, Hsia J, Kinney HC, Mandell F, McClain M, Randall B, Habbe D, Wilson H, Willinger M. Risk factors for sudden infant death syndrome among northern plains Indians. JAMA. 2002 Dec 4;288(21):2717-23. doi: 10.1001/jama.288.21.2717. PMID 12460095
- [Background] Heil SH, Jones HE, Arria A, Kaltenbach K, Coyle M, Fischer G, Stine S, Selby P, Martin PR. Unintended pregnancy in opioid-abusing women. J Subst Abuse Treat. 2011 Mar;40(2):199-202. doi: 10.1016/j.jsat.2010.08.011. Epub 2010 Oct 30. PMID 21036512
- [Background] Ko JY, Wolicki S, Barfield WD, Patrick SW, Broussard CS, Yonkers KA, Naimon R, Iskander J. CDC Grand Rounds: Public Health Strategies to Prevent Neonatal Abstinence Syndrome. MMWR Morb Mortal Wkly Rep. 2017 Mar 10;66(9):242-245. doi: 10.15585/mmwr.mm6609a2. PMID 28278146
- [Background] National Academies of Sciences, Engineering, and Medicine; Health and Medicine Division; Board on Population Health and Public Health Practice; Committee on the Examination of the Integration of Opioid and Infectious Disease Prevention Efforts in Select Programs. Opportunities to Improve Opioid Use Disorder and Infectious Disease Services: Integrating Responses to a Dual Epidemic. Washington (DC): National Academies Press (US); 2020 Jan 23. Available from http://www.ncbi.nlm.nih.gov/books/NBK555809/ PMID 32293827
- [Background] Terplan M, Lawental M, Connah MB, Martin CE. Reproductive Health Needs Among Substance Use Disorder Treatment Clients. J Addict Med. 2016 Jan-Feb;10(1):20-5. doi: 10.1097/ADM.0000000000000175. PMID 26690290
- [Background] Cornford CS, Close HJ, Bray R, Beere D, Mason JM. Contraceptive use and pregnancy outcomes among opioid drug-using women: a retrospective cohort study. PLoS One. 2015 Mar 4;10(3):e0116231. doi: 10.1371/journal.pone.0116231. eCollection 2015. PMID 25739018
- [Background] Stanhope TJ, Gill LA, Rose C. Chronic opioid use during pregnancy: maternal and fetal implications. Clin Perinatol. 2013 Sep;40(3):337-50. doi: 10.1016/j.clp.2013.05.015. Epub 2013 Jul 4. PMID 23972743
- [Background] Kellogg A, Rose CH, Harms RH, Watson WJ. Current trends in narcotic use in pregnancy and neonatal outcomes. Am J Obstet Gynecol. 2011 Mar;204(3):259.e1-4. doi: 10.1016/j.ajog.2010.12.050. PMID 21376165
- [Background] Pinedo M. Help seeking behaviors of Latinos with substance use disorders who perceive a need for treatment: Substance abuse versus mental health treatment services. J Subst Abuse Treat. 2020 Feb;109:41-45. doi: 10.1016/j.jsat.2019.11.006. Epub 2019 Nov 14. PMID 31856949
- [Background] Hadland SE, Copelas SH, Harris SK. Trajectories of Substance Use Frequency among Adolescents Seen in Primary Care: Implications for Screening. J Pediatr. 2017 May;184:178-185. doi: 10.1016/j.jpeds.2017.01.033. Epub 2017 Feb 10. PMID 28196680
- [Background] Chavez LJ, Kelleher KJ, Matson SC, Wickizer TM, Chisolm DJ. Mental Health and Substance Use Care Among Young Adults Before and After Affordable Care Act (ACA) Implementation: A Rural and Urban Comparison. J Rural Health. 2018 Dec;34(1):42-47. doi: 10.1111/jrh.12258. Epub 2017 Jul 7. PMID 28685885
- [Background] Robbins C, Boulet SL, Morgan I, D'Angelo DV, Zapata LB, Morrow B, Sharma A, Kroelinger CD. Disparities in Preconception Health Indicators - Behavioral Risk Factor Surveillance System, 2013-2015, and Pregnancy Risk Assessment Monitoring System, 2013-2014. MMWR Surveill Summ. 2018 Jan 19;67(1):1-16. doi: 10.15585/mmwr.ss6701a1. PMID 29346340
- [Background] Hayes DK, Robbins CL, Ko JY. Trends in Selected Chronic Conditions and Related Risk Factors Among Women of Reproductive Age: Behavioral Risk Factor Surveillance System, 2011-2017. J Womens Health (Larchmt). 2020 Dec;29(12):1576-1585. doi: 10.1089/jwh.2019.8275. Epub 2020 May 22. PMID 32456604
- [Background] Hall KS, Samari G, Garbers S, Casey SE, Diallo DD, Orcutt M, Moresky RT, Martinez ME, McGovern T. Centring sexual and reproductive health and justice in the global COVID-19 response. Lancet. 2020 Apr 11;395(10231):1175-1177. doi: 10.1016/S0140-6736(20)30801-1. No abstract available. PMID 32278371
- [Background] ACOG Committee on Health Care for Underserved Women; American Society of Addiction Medicine. ACOG Committee Opinion No. 524: Opioid abuse, dependence, and addiction in pregnancy. Obstet Gynecol. 2012 May;119(5):1070-6. doi: 10.1097/AOG.0b013e318256496e. PMID 22525931
- [Background] Frost JJ, Gold RB, Bucek A. Specialized family planning clinics in the United States: why women choose them and their role in meeting women's health care needs. Womens Health Issues. 2012 Nov-Dec;22(6):e519-25. doi: 10.1016/j.whi.2012.09.002. PMID 23122212
- [Background] Hall KS, Harris LH, Dalton VK. Women's Preferred Sources for Primary and Mental Health Care: Implications for Reproductive Health Providers. Womens Health Issues. 2017 Mar-Apr;27(2):196-205. doi: 10.1016/j.whi.2016.09.014. Epub 2016 Nov 4. PMID 27825589
- [Background] Friedmann PD, McCullough D, Chin MH, Saitz R. Screening and intervention for alcohol problems. A national survey of primary care physicians and psychiatrists. J Gen Intern Med. 2000 Feb;15(2):84-91. doi: 10.1046/j.1525-1497.2000.03379.x. PMID 10672110
- [Background] Wright TE, Terplan M, Ondersma SJ, Boyce C, Yonkers K, Chang G, Creanga AA. The role of screening, brief intervention, and referral to treatment in the perinatal period. Am J Obstet Gynecol. 2016 Nov;215(5):539-547. doi: 10.1016/j.ajog.2016.06.038. Epub 2016 Jul 1. PMID 27373599
- [Background] Rahm AK, Boggs JM, Martin C, Price DW, Beck A, Backer TE, Dearing JW. Facilitators and Barriers to Implementing Screening, Brief Intervention, and Referral to Treatment (SBIRT) in Primary Care in Integrated Health Care Settings. Subst Abus. 2015;36(3):281-8. doi: 10.1080/08897077.2014.951140. Epub 2014 Aug 15. PMID 25127073
- [Background] Hettema J, Cockrell S, Russo J, Corder-Mabe J, Yowell-Many A, Chisholm C, Ingersoll K. Missed Opportunities: Screening and Brief Intervention for Risky Alcohol Use in Women's Health Settings. J Womens Health (Larchmt). 2015 Aug;24(8):648-54. doi: 10.1089/jwh.2014.4961. Epub 2015 Jul 31. PMID 26230758
- [Background] Goldstein KM, Zullig LL, Dedert EA, Alishahi Tabriz A, Brearly TW, Raitz G, Sata SS, Whited JD, Bosworth HB, Gordon AM, Nagi A, Williams JW Jr, Gierisch JM. Telehealth Interventions Designed for Women: an Evidence Map. J Gen Intern Med. 2018 Dec;33(12):2191-2200. doi: 10.1007/s11606-018-4655-8. Epub 2018 Oct 3. PMID 30284173
- [Background] Boudreaux ED, Haskins B, Harralson T, Bernstein E. The remote brief intervention and referral to treatment model: Development, functionality, acceptability, and feasibility. Drug Alcohol Depend. 2015 Oct 1;155:236-42. doi: 10.1016/j.drugalcdep.2015.07.014. Epub 2015 Jul 23. PMID 26297297
- [Background] Becker SJ, Murphy CM, Hartzler B, Rash CJ, Janssen T, Roosa M, Madden LM, Garner BR. Project MIMIC (Maximizing Implementation of Motivational Incentives in Clinics): A cluster-randomized type 3 hybrid effectiveness-implementation trial. Addict Sci Clin Pract. 2021 Oct 12;16(1):61. doi: 10.1186/s13722-021-00268-0. PMID 34635178
- [Background] Garner BR, Zehner M, Roosa MR, Martino S, Gotham HJ, Ball EL, Stilen P, Speck K, Vandersloot D, Rieckmann TR, Chaple M, Martin EG, Kaiser D, Ford JH 2nd. Testing the implementation and sustainment facilitation (ISF) strategy as an effective adjunct to the Addiction Technology Transfer Center (ATTC) strategy: study protocol for a cluster randomized trial. Addict Sci Clin Pract. 2017 Nov 17;12(1):32. doi: 10.1186/s13722-017-0096-7. PMID 29149909
- [Background] Garner BR, Gotham HJ, Chaple M, Martino S, Ford Ii JH, Roosa MR, Speck KJ, Vandersloot D, Bradshaw M, Ball EL, Toro AK, Griggs C, Tueller SJ. The implementation and sustainment facilitation strategy improved implementation effectiveness and intervention effectiveness: Results from a cluster-randomized, type 2 hybrid trial. Implement Res Pract. 2020 Jan-Dec;1:2633489520948073. doi: 10.1177/2633489520948073. Epub 2020 Sep 7. PMID 36189179
- [Background] Gotham HJ, Wilson K, Carlson K, Rodriguez G, Kuofie A, Witt J. Implementing Substance Use Screening in Family Planning. J Nurse Pract. 2019;15(4):306-310.